CLINICAL TRIAL: NCT03058055
Title: Brain Exercises for Synaptic Plasticity: the BEST Study
Brief Title: Brain Exercises for Synaptic Plasticity
Acronym: BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Gregory Jicha, 323-5550, M.D., Ph.D., Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEST
Record Dates: First submitted 2017-02-12; First posted 2017-02-20 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Cognitive Change

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Usual lifestyle activities
  Interventions: Behavioral: Placebo
- Origami (Experimental): Origami lessons (one hour/week) with daily take home Origami activities to complete
  Interventions: Behavioral: Origami
- Reading (Experimental): Daily reading (out loud into a voice recorder) for one hour
  Interventions: Behavioral: Reading

INTERVENTIONS:
Behavioral: Placebo — The placebo group will have unstructured lifestyle activities (normal lifestyle activities without restraint).
  Arms: Placebo
Behavioral: Origami — Origami lessons (one hour/week) with daily take home Origami activities to complete
  Arms: Origami
Behavioral: Reading — Book club that includes weekly one hour meetings and daily reading assignments
  Arms: Reading

SUMMARY:
The BEST study will investigate the feasibility of cognitive interventions in a randomized, placebo-controlled, clinical trial. The investigators will recruit 45 cognitively normal subjects and engage them in one of three cohorts over an 8 week period, including active reading vs. origami study arms and a placebo group without structured cognitive intervention.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled study investigating the practical implementation and conduct of two cognitive interventions in non-demented subjects. Subjects will be randomized 1:1:1 into three groups including: 1) a Book club that includes weekly one hour meetings and daily reading assignments, 2) Origami lessons (one hour/week) with daily take home Origami activities to complete, and 3) a placebo group with unstructured lifestyle activities (normal lifestyle activities without restraint).

ELIGIBILITY:
Inclusion Criteria:

* Non demented community dwelling elders

Exclusion Criteria:

* Unable to perform the reading or origami tasks for any reason

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
MOCA | 8 weeks
  The Montreal Cognitive Assessment (MOCA) measures general cognitive function
FCSRT | 8 weeks
  The Free and Cued Selective Reminding Test (FCSRT) measures memory function.

SECONDARY OUTCOMES:
Adherence to protocol | 8 weeks
  Objective measures of weekly time devoted to cognitive training activities
Electroencephalogram | 8 weeks
  resting state electroencephalogram pattern
Evoked Related Potential | 8 weeks
  Evoked Related Potential P300 using the Bluegrass memory task

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Jicha, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Sander's Brown Center on Aging, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No